CLINICAL TRIAL: NCT00912392
Title: Etoposide-Carboplatin (EC) Versus EC Plus Endostar in Patients With Extensive Disease Small Cell Lung Cancer (ED-SCLC): Randomized, Open Label, Placebo-controlled, Multicentre Study
Brief Title: Etoposide-Carboplatin Alone or With Endostar for Extensive Disease Small Cell Lung Cancer (ED-SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Simcere-Medgenn Bio-pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-69
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — endostar protein; EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoposide-Carboplatin with Endostar (Experimental): Endostar® 7.5mg/m2 on day 1 to day 14, etoposide 60 mg/m2 on day 1 to day 5 and carboplatin AUC 5 on day 1.
  Interventions: Drug: Endostar; Drug: Etoposide-Carboplatin
- Etoposide-Carboplatin (Active Comparator): Etoposide 60 mg/m2 on day 1 to day 5 and carboplatin AUC 5 on day 1.
  Interventions: Drug: Etoposide-Carboplatin

INTERVENTIONS:
Drug: Endostar — Endostar® 7.5mg/m2 on day 1 to day 14
  Arms: Etoposide-Carboplatin with Endostar
Drug: Etoposide-Carboplatin — Etoposide 60 mg/m2 on day 1 to day 5 and carboplatin AUC 5 on day 1.

SUMMARY:
Background:

The effect of existing treatment modalities of extensive disease small-cell lung cancer (ED-SCLC) is unsatisfactory. Progress of new strategies including more efficient therapy is wanted. Endostar® (Rh-endostatin Injection) may have anti-tumor activity by against vascular endothelial growth factor for initial treatment. This study was designed to evaluate the safety and efficacy of Endostar® combined with etoposide-carboplatin (EC) chemotherapy in patients with ED-SCLC seeking for more effective treatment.

DETAILED DESCRIPTION:
Methods:

In this randomized, open label, placebo-controlled, multicentre trial, 120 patients are planned to be enrolled at random into 2 arms(1:1) from 10 centers between June 2009 and June 2011. The leader units are Shanghai Chest Hospital Affiliated to Shanghai Jiao-Tong University. Main eligibility criteria are histological or cytological diagnosis of ED-SCLC, with an age of 18-75 years. All eligible patients receive etoposide-carboplatin (EC) alone or with endostar® for 4-6 cycles (21 days for 1 cycle). In arm1 patients receive endostar® 7.5mg/m2 on day 1 to day 14, etoposide 60 mg/m2 on day 1 to day 5 and carboplatin AUC 5 on day 1. In arm2 patients receive etoposide 60 mg/m2 on day 1 to day 5 and carboplatin AUC 5 on day 1.

Primary endpoint: progress free survival (PFS).

Secondary endpoint: progress free survival at 6 months, overall survival (OS), objective response rate (ORR), clinical benefit rate (CBR), Response duration, time to progression(TTP) and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed SCLC;
* Age of 18-75 years;
* Life expectancy > 3 months;
* Adequate hematologic, renal, and hepatic function;
* ECOG PS 0-2;

Exclusion Criteria:

* Brain metastases;
* Clinically significant cardiovascular disease;
* Presence of hepatic and renal dysfunction;
* Evidence of bleeding diathesis or coagulopathy
* Pregnant or lactating woman;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Oct-30-2012

SECONDARY OUTCOMES:
Progression free survival | at 6 months
Overall survival (OS) | Oct-30-2012
Objective response rate (ORR) | Oct-30-2012
Clinical benefit rate (CBR) | Oct-30-2012
Response duration | Oct-30-2012
Time to progression(TTP) | Oct-30-2012
Quality of life (QOL) | Oct-30-2012

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Dr., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China